CLINICAL TRIAL: NCT00648232
Title: HIV Counseling and Testing and Linkage to Care in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas J. Coates, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH077512 (NIH); R01MH077512 (NIH); DABHR 9A-ASGA
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Prevention; VCT; Voluntary Counseling and Testing
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A (Experimental): Participants will receive voluntary brief HIV counseling and testing plus enhanced linkage to care.
  Interventions: Behavioral: Voluntary brief HIV counseling and testing; Behavioral: Enhanced linkage to care
- B (Experimental): Participants will receive voluntary brief HIV counseling and testing plus routine referral to care.
  Interventions: Behavioral: Voluntary brief HIV counseling and testing; Behavioral: Routine referral to care
- C (Experimental): Participants will receive voluntary longer, more detailed HIV counseling and testing plus enhanced linkage to care.
  Interventions: Behavioral: Voluntary longer, more detailed HIV counseling and testing; Behavioral: Enhanced linkage to care
- D (Experimental): Participants will receive voluntary longer, more detailed HIV counseling and testing plus routine referral to care.
  Interventions: Behavioral: Voluntary longer, more detailed HIV counseling and testing; Behavioral: Routine referral to care
- E (Active Comparator): Participants who are found to be healthy will receive voluntary brief HIV counseling and testing only.
  Interventions: Behavioral: Voluntary brief HIV counseling and testing
- F (Active Comparator): Participants who are found to be healthy will receive voluntary longer, more detailed HIV counseling and testing only.
  Interventions: Behavioral: Voluntary longer, more detailed HIV counseling and testing

INTERVENTIONS:
Behavioral: Voluntary brief HIV counseling and testing — Participants will receive 10 to 15 minutes of pretest counseling on the importance of HIV testing and on available services for people infected with HIV. After pretest counseling, participants will undergo a blood draw for HIV testing. Participants will receive test results and additional counseling 1 hour after the blood sample is drawn.
  Arms: A; B; E
Behavioral: Voluntary longer, more detailed HIV counseling and testing — Participants will receive 45 to 60 minutes of pretest counseling on general HIV/AIDS information and testing for HIV. After pretest counseling, participants will undergo a blood draw for HIV testing. Participants will receive test results and additional counseling 1 hour after the blood sample is drawn.
  Arms: C; D; F
Behavioral: Enhanced linkage to care — Participants will be provided with more detailed counseling on how to access HIV services, will be introduced to a specific HIV clinic, and will be given a list of other HIV services available in the area. After leaving the hospital, participants will receive reminder telephone calls 1 week before their scheduled visits at the HIV clinics.
  Arms: A; C
Behavioral: Routine referral to care — Participants will be provided with information on the importance of receiving HIV care and will be given a list of available HIV area services.
  Arms: B; D

SUMMARY:
This study will compare the effectiveness of brief versus detailed HIV counseling sessions, paired with referrals to either HIV-specific medical care or usual care, in reducing HIV risk behavior and in increasing treatment adherence in Uganda.

DETAILED DESCRIPTION:
HIV is a virus that can lead to acquired immunodeficiency syndrome (AIDS), a disease that breaks down the immune system and allows for entry of life-threatening secondary infections. HIV is a major global health concern, with countries in Africa undergoing a severe HIV/AIDS crisis. The number of new cases of HIV infection in Africa continues to rise, making disease prevention methods imperative. Important to the prevention process are early testing, educational counseling on HIV and how to reduce sexual-risk behavior, and connecting people with HIV infection to services that offer medical treatment and social support. However, the most effective strategy for fully integrating HIV counseling, testing, and medical care access is not known. This study will compare the effectiveness of brief versus detailed HIV counseling sessions, paired with either referrals to HIV-specific medical care or usual care, in reducing HIV risk behavior and in increasing treatment adherence in Uganda.

Participation in this study will last 12 months. All participants will undergo an initial interview to obtain basic information on previous HIV testing and status. Participants will then be assigned randomly to receive a brief or more detailed counseling session given before and after HIV testing. Participants assigned to the brief counseling session will receive 10 to 15 minutes of pretest counseling on the importance of HIV testing and available services for people infected with HIV. Participants assigned to the detailed counseling session will receive 45 to 60 minutes of pretest counseling on general HIV/AIDS information and testing for HIV. After pretest counseling, participants in both groups will undergo a blood draw for HIV testing. All participants will receive test results and additional counseling 1 hour after the blood sample is drawn.

Participants who are found to be infected with HIV will be assigned randomly to receive enhanced referrals to HIV-specific medical care or referrals to usual care. Participants receiving the enhanced referrals will be provided with more detailed counseling on how to access HIV services, will be introduced to a specific HIV clinic, and will be given a list of other HIV services available in the area. After leaving the hospital, participants will receive reminder telephone calls 1 week before their first scheduled visits at the HIV clinics. Participants receiving referrals to usual care will be provided with information on the importance of receiving HIV care and will be given a list of available HIV area services. At Months 3, 6, 9, and 12, participants in both groups will be interviewed about contact information, overall health, current medications, sexual history, health services utilized, and any repeat HIV tests. Participants who are not infected with HIV may be randomly selected to undergo the same follow-up interviews as the HIV infected participants.

ELIGIBILITY:
Inclusion Criteria:

* Willing to receive HIV test results
* Willing to provide adequate contact information
* Possesses sufficient cognitive ability to provide informed consent and participate in the interventions, as determined subjectively by the Regulatory Coordinator (patient with altered mental status or who is otherwise too ill to participate in the consent process will be excluded)
* Planned local residence over the next year after study entry (within a reasonable distance; approximate radius of 25 km of Kampala city center)
* Fluent in Luganda or English

Exclusion Criteria:

* Self-reported HIV-infected serostatus (defined as ever receiving an HIV-positive test result)
* Self-reported HIV test within the 12 months before study entry
* Any condition that, in the opinion of the study staff, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3415 (Actual)
Dates: Start 2008-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Reduction in HIV risk behavior among inpatients after discharge | Measured at Months 3, 6, 9, and 12
Receipt of opportunistic infection (OI) prophylaxis, adherence to antiretroviral therapy (ART), and reduction in mortality | Measured at Months 3, 6, 9, and 12

SECONDARY OUTCOMES:
Number of infections averted per patient randomized to each of the four intervention strategies | Measured at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Coates, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Makerere University/Mulago Teaching Hospital, Uganda, Kampala, Uganda

REFERENCES:
- [Derived] Wanyenze RK, Kamya MR, Fatch R, Mayanja-Kizza H, Baveewo S, Szekeres G, Bangsberg DR, Coates T, Hahn JA. Abbreviated HIV counselling and testing and enhanced referral to care in Uganda: a factorial randomised controlled trial. Lancet Glob Health. 2013 Sep;1(3):e137-45. doi: 10.1016/S2214-109X(13)70067-6. Epub 2013 Aug 23. PMID 25104262